CLINICAL TRIAL: NCT04263220
Title: Testing the Effectiveness and Safety of a New Prototype of a Passive Industrial Exoskeleton for Back Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Scientific Institution "Izmerov Research Institute of Occupational Health" (Other)
Responsible Party: Principal Investigator, Andrey Mikhailovich Geregey, Head of the Laboratory of Personal Protective Equipment and Industrial Exoskeletons Andrey Geregey, Federal State Budgetary Scientific Institution "Izmerov Research Institute of Occupational Health"
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PPE-01
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Prevention of Diseases of the Musculoskeletal System
Keywords: industrial exoskeleton; exoskeleton; passive industrial exoskeleton

STUDY DESIGN:
Intervention Model Description: Randomized counterbalanced cross-over design
Who Masked: Participant
Masking Description: Blinding is not possible in this testing set-up, participants however are not informed about the exact purpose of the tests and which exoskeleton is a prototype and which exoskeleton is a commercially available exoskeleton
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prototype exoskeleon 1 (Experimental): The experimental trial will be performed with the prototype exoskeleton
  Interventions: Device: Industrial passive exoskeleton with a specific value of the torque of the spring for supporting the back
- Prototype exoskeleon 2 (Experimental): The experimental trial will be performed with the prototype exoskeleton
  Interventions: Device: Industrial passive exoskeleton with a specific value of the torque of the spring for supporting the back
- No exoskeleton (Experimental): The experimental protocol will be performed without exoskeleton.
  Interventions: Other: protocol will be performed without exoskeleton

INTERVENTIONS:
Device: Industrial passive exoskeleton with a specific value of the torque of the spring for supporting the back — Both exoskeleton types are passive exoskeletons for supporting the back. The goal is to compare the human response to the simulated industrial tasks between the different exoskeleton conditions
  Arms: Prototype exoskeleon 1; Prototype exoskeleon 2
Other: protocol will be performed without exoskeleton — protocol will be performed without exoskeleton
  Arms: No exoskeleton

SUMMARY:
This research will provide data on evaluation of the effectiveness and safety of using a passive exoskeleton designed to reduce the negative impact of static and dynamic loads associated with body tilts, lifting and holding weights on the musculoskeletal system of workers. To evaluate a passive industrial exoskeleton for back support, a protocol was developed in which individual production operations will be modeled.

This research will recruit 9 valunteers. During a 4-hour laboratory visit, each subject will perform three identical experimental tests: one test without an exoskeleton and two tests using two different modifications of the exoskeleton prototype. To avoid sequence bias, the test order will be randomized (balanced). Two types of labor operations will be simulated. One operation will consist in lifting the load, which is 20% of the volunteer's body weight, from a height of 14 cm to a surface with a height of 70 cm, the frequency of lifting is 1 time in 30 seconds. The second operation is holding a cargo weighing 5 kg in a forced working position (tilt of the body more than 30 °) for 1 minute, after which rest will follow for 1 minute, and then the work will be repeated. Both types of work will be performed for 105 minutes, then a break of 15 minutes, then 105 minutes of work. Heart rate, blood pressure, ECG (Custo) will be monitored. An ergospirometric device (Metamax) will be used to collect muscle activity data (Trust-M, Myoton), inertial sensors (Trust-M) will be used to evaluate the biomechanics of movements. In addition, questionnaires will be filled out for a subjective assessment of the use of exoskeleton prototypes (local discomfort scale, exoskeleton properties assessment questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals (based on medical screening)

Exclusion Criteria:

* musculoskeletal system diseases
* musculoskeletal injuries
* health deviations at the time of the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Heart rate | 6 hours
  A Polar H10 heart rate monitor (Polar Electro, Finland) will carry all items during the entire research
Blood pressure | 6 hours
  A Custo med blood pressure monitor will be used by all subjects throughout the study
Range of motion in large joints of the upper, lower limbs and spine | 1 hour
  Inertial sensors will be mounted on the body of the volunteer. The amplitude of the moving in the shoulder, elbow, hip, knee joints and in the thoracolumbar spine is determined. Flexion and extension, abduction and adduction, rotation are performed.
Metabolic cost of ergospirometric testing | 4 hours
  A Metamax 3B instrument (Cortex, Germany) will be used to measure a metabolic cost during all labor activities, 4 hours.
Surface electromyography | 1.5 hours
  Trust-M sensors with electrodes will be used to collect electromyographic data in accordance with the SENIAM recommendations. The muscles that will be monitored, the muscles of the arms, legs and back, which account for the maximum load. The locations of the sensors will be prepared by shaving, abrasion with sandpaper, and alcohol cleaning. The average amplitude of the EMG spectrum will be collected. The recording will be carried out at rest, standing before and after work, as well as outside work in the voltage position without exoskeleton and with it.
Myotonometry | 1.5 hours
  Myotonometry will be performed with a Myoton Pro device. Parameters of the certain muscles, which get the maximum load, will be measured at rest standing before and after work, as well as outside work in a stress position without an exoskeleton and with it.
Local Comfort Rating Scale | 1 hour
  This questionnaire is for assessing the duration of maintaining a working posture without discomfort, fixing their appearance, as well as the nature of these sensations. Points can vary from 1 to 10, where 1 is the absence of pain, 10 is unbearable pain.

SECONDARY OUTCOMES:
Exoskeleton parameter evaluation form | 30 minutes
  The questionnaire contains questions related to the operational, ergonomic and aesthetic characteristics of the exoskeleton. The assessment will be carried out in points on a scale from -2 to +2.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Scientific Institution Izmerov Research Institute of Occupational Health, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No